CLINICAL TRIAL: NCT00467636
Title: Influence of Insulin Therapy in Patients Admitted to Hospital With Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Insulin Therapy in Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting (early discharge scheme initiated)
Sponsor: The Royal Bournemouth Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Professor David Kerr, Royal Bournemouth Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COPD1
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hyperglycemia
Keywords: Chronic Obstructive Pulmonary Disease; Corticosteroid induced hyperglycaemia; Insulin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperglycemia; Insulin Resistance | interventions — Blood Glucose; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Glulisine (Experimental): Blood glucose monitoring and treatment of hyperglycaemia with insulin. Insulin to be with-held if pre meal blood glucose < 4 mmol/l.
  Interventions: Drug: Insulin Glulisine
- 2 (Active Comparator): Blood glucose monitoring for comparison with treatment arm (1)
  Interventions: Procedure: Blood glucose monitoring

INTERVENTIONS:
Procedure: Blood glucose monitoring — Regular pre and post meal blood glucose monitoring.
  Arms: 2
Drug: Insulin Glulisine — Sub cutaneous injection given twice daily for 3 days. Dosage titrated to body mass index and body weight (BMI < 30 = 0.1 unit/kg. BMI > 30 = 0.2 unit/kg)
  Other Names: Apidra
  Arms: Insulin Glulisine

SUMMARY:
The purpose of this study is to determine the effect of preventing hyperglycaemia in patients admitted to hospital with acute exacerbations of chronic pulmonary disease.

DETAILED DESCRIPTION:
Hyperglycaemia is associated with increased morbidity and mortality in patients admitted to hospital with acute critical illness, myocardial infarction and stroke. Moreover patients with hyperglycaemia have a significantly longer hospital stay, higher rates of ICU admission, increased in-hospital mortality and are more likely to require transfer to a nursing home. Recently, interventional studies have linked reversal of hyperglycaemia to better clinical outcomes especially in acute myocardial infarction, cardiac surgery and in critically ill patients.

In England and Wales, it is estimated that the number of people with COPD is approaching 1.5 million. The morbidity and economic costs associated with the condition are extremely high with approximately 10% of all acute medical admissions caused by exacerbations of the underlying condition. As a corollary about 15% of patients with COPD need admission to hospital each year.

Acute hyperglycaemia is common among patients admitted with acute exacerbations of COPD. The reasons for this are likely to be multi-factorial including an association between COPD and increased risk of developing diabetes at least in women, the elderly nature of the two populations and the use of glucocorticoids which markedly increases the risk of hyperglycaemia. Admission hyperglycaemia (>11 mmol/l) also appears to predict increased morbidity for patients with COPD admitted to intensive care.

The trial will be a randomised trial of comparison of usual treatment vs intensive insulin treatment for patients with COPD who may or may not have diabetes. Patients will take part in the trial for the first 5 days during their hospital stay.

ELIGIBILITY:
Inclusion criteria

* Patients who are NOT diabetic, admitted with COPD who are likely to be prescribed corticosteroids as part of usual care with an admission glucose level (before steroids) between 6.1 and 11.1 mmol/l.

Exclusion criteria:

* Patients with diabetes mellitus
* Patients who are nil by mouth.
* Patients with severe co-morbid disease with an anticipated life expectancy of < 6 months.
* Patients who are unable to provide informed consent.
* Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Rate of re-admission to hospital within 90 days. | 90 days after discharged from hospital

SECONDARY OUTCOMES:
Length of stay | oct 2009
In-patient mortality | look at cause death. for statistical purpose oct 2009
Spirometry at baseline, day 3 and prior to discharge | oct 2009
Achieved glucose levels | oct 2009
Hypoglycaemic events (<4 mmol/l with or without symptoms) | instigate hypoglycaemia protocol at time. for statistical purpose oct 2009.
Frequency of positive sputum cultures | oct 2009
Change in CRP and IL-6 levels between baseline and day 5 | oct 2009

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, MD, Principal Investigator — Royal Bournemouth Hospital NHS Trust
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom